CLINICAL TRIAL: NCT03505892
Title: A Real-world, Prospective, Observational Study to Investigate the Clinical REsponses in Ankylosing Spondylitis Patients on Adalimumab Therapy in Taiwan (EAST)
Brief Title: A Study to Investigate the Clinical REsponses in Ankylosing Spondylitis Patients on Adalimumab Therapy in Taiwan (EAST)
Acronym: EAST
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P16-326
Record Dates: First submitted 2018-03-30; First posted 2018-04-23 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Ankylosing Spondylitis (AS)
Keywords: Ankylosing Spondylitis (AS); Adaliumumab; Humira
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants receiving adalimumab: Participants with AS receiving adalimumab

SUMMARY:
The objectives of this prospective observational study is to explore 1-year clinical response via both Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) and Ankylosing Spondylitis Disease Activity Score (ASDAS) after initiation of adalimumab therapy in AS patients from routine clinical practices in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Participants with confirmed AS.
* Participant will start adalimumab as treatment
* Participant must provide the written authorization form and agree to provide personal and/or health data prior to the entry into the study.

Exclusion Criteria:

* Participant has been treated with any investigational drug or biologic within a minimum of 30 days or five half-lives (whichever is longer) of the drug prior to the Baseline Visit.
* Participants who fulfill any of the contraindications as per Humira label in Taiwan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Ankylosing Spondylitis (AS) after the initiation of adalimumab therapy in the real-world practices in Taiwan.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Percentage of participants that achieve 50% improvement of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at Week 24 | 24 Weeks after initiation of Humira therapy
  This accounts for participants achieving 50% improvement in BASDAI.

SECONDARY OUTCOMES:
Percentages of participants who achieve major improvement of Ankylosing Spondylitis Disease Activity Score (ASDAS) at Week 24 | 24 Weeks after initiation of Humira therapy
  The ASDAS tool is a self-administered questionnaire plus an objective laboratory evaluation.
Percentages of participants who achieve clinically important improvement of Ankylosing Spondylitis Disease Activity Score (ASDAS) at Week 24 | 24 Weeks after initiation of Humira therapy
  The ASDAS tool is a self-administered questionnaire plus an objective laboratory evaluation.
Percentage of participants that achieve 50% improvement of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Every 12 weeks' follow-up after initiation of Humira therapy (approximately up to 58 weeks)
  This accounts for participants achieving 50% improvement in BASDAI.
Percentages of participants who achieve clinically important improvement of Ankylosing Spondylitis Disease Activity Score (ASDAS) | Every 12 weeks' follow-up after initiation of Humira therapy (approximately up to 58 weeks)
  The ASDAS tool is a self-administered questionnaire plus an objective laboratory evaluation.
Percentages of participants who achieve major improvement of Ankylosing Spondylitis Disease Activity Score (ASDAS) | Every 12 weeks' follow-up after initiation of Humira therapy (approximately up to 58 weeks)
  The ASDAS tool is a self-administered questionnaire plus an objective laboratory evaluation.
Percentages of participants whose disease activity states are inactive per ASDAS score | At Week 0 (Baseline) and every 12 weeks' follow-up after initiation of Humira therapy (approximately up to 58 weeks)
  The ASDAS tool is a self-administered questionnaire plus an objective laboratory evaluation.
Percentages of participants whose disease activity states are moderate per ASDAS score | At Week 0 (Baseline) and every 12 weeks' follow-up after initiation of Humira therapy (approximately up to 58 weeks)
  The ASDAS tool is a self-administered questionnaire plus an objective laboratory evaluation.
Changes of the frequency of overall extra-articular manifestations (EAM) of interest | At Week 0 (Baseline) and every 12 weeks' follow-up after initiation of Humira therapy (approximately up to 58 weeks)
  The change of the frequency of overall extra-articular manifestations (EAM) will be assessed.
Changes of the respective frequency of each EAM | At Week 0 (Baseline) and every 12 weeks' follow-up after initiation of Humira therapy (approximately up to 58 weeks)
  The changes of the respective frequency of each EAM will be assessed.
Changes in the percentage of participants who have enthesitis of the plantar fascia or Achilles tendon | At Week 0 (Baseline) and every 12 weeks' follow-up after initiation of Humira therapy (approximately up to 58 weeks)
  The change in the percentage of participants who have enthesitis of the plantar fascia or Achilles tendon will be assessed.
Change in Maastricht Ankylosing Spondylitis Enthesitis Score (MASES) | At Week 0 (Baseline) and every 12 weeks' follow-up after initiation of Humira therapy (approximately up to 58 weeks)
  The change in MASES score will be assessed.
Change in Tender Joint Counts (TJC) | At Week 0 (Baseline) and every 12 weeks' follow-up after initiation of Humira therapy (approximately up to 58 weeks)
  The change of TJC (0-46), in participants who had peripheral arthritis (≥1 swollen joint) at baseline will be assessed.
Change in Swollen Joint Counts (SJC) | At Week 0 (Baseline) and every 12 weeks' follow-up after initiation of Humira therapy (approximately up to 58 weeks)
  The change of SJC (0-44), in participants who had peripheral arthritis (≥1 swollen joint) at baseline will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Hualien Tzuchi Hospital, The Buddhist Tzuchi Medical Foundation, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=P16-326#additional-resources-section